CLINICAL TRIAL: NCT01895309
Title: A Randomised, Double-blind, Parallel Group, Multicentre Clinical Study to Evaluate the Efficacy, Safety, Pharmacokinetics and Immunogenicity of SB4 Compared to Enbrel® in Subjects With Moderate to Severe Rheumatoid Arthritis Despite Methotrexate Therapy
Brief Title: A Study Comparing SB4 to Enbrel® in Subjects With Moderate to Severe Rheumatoid Arthritis Despite Methotrexate Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB4-G31-RA
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Results first posted 2016-08-29 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2015-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Etanercept; Biosimilar
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SB4 (proposed biosimilar to etanercept) (Experimental): SB4 50 mg/week via subcutaneous injection
  Interventions: Drug: SB4 (proposed biosimilar to etanercept)
- Enbrel (etanercept) (Active Comparator): Enbrel 50 mg/week via subcutaneous injection
  Interventions: Drug: Enbrel (etanercept)

INTERVENTIONS:
Drug: Enbrel (etanercept)
  Arms: Enbrel (etanercept)
Drug: SB4 (proposed biosimilar to etanercept)
  Arms: SB4 (proposed biosimilar to etanercept)

SUMMARY:
This is a randomized, double-blind, parallel group, multicentre clinical study to evaluate the efficacy, safety, pharmacokinetics and immunogenicity of SB4 compared to Enbrel in subjects with moderate to severe Rheumatoid Arthritis (RA) despite Methotrexate (MTX) therapy. In some countries, after 52 weeks of treatment with either SB4 or Enbrel, subjects will be enrolled into an open label extension period. Subjects will receive SB4 for an additional 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as having RA according to the revised 1987 ACR criteria for at least 6 months but not exceeding 15 years prior to Screening
* Have moderate to severe active disease despite MTX therapy defined as having more than or equal to six swollen joints and more than or equal to six tender joints and either erythrocyte sedimentation rate (ESR, Westergren) ≥ 28 mm/h or serum C-reactive protein ≥ 1.0 mg/dL
* Must have been treated with MTX for at least 6 months prior to Randomisation and on a stable dose of MTX 10-25 mg/week given at least 4 weeks prior to Screening
* Female subjects who are not pregnant or nursing at Screening and who are not planning to become pregnant from Screening until 2 months after the last dose of investigational product

Exclusion Criteria:

* Have been treated previously with any biological agents including any tumour necrosis factor inhibitor
* Have a known hypersensitivity to human immunoglobulin proteins or other components of Enbrel or SB4
* Have a positive serological test for hepatitis B or hepatitis C or have a known history of infection with human immunodeficiency virus
* Have a current diagnosis of active tuberculosis
* Have had a serious infection or have been treated with intravenous antibiotics for an infection within 8 weeks or oral antibiotics within 2 weeks prior to Randomisation.
* Have any of the following conditions

  1. Other inflammatory or rheumatic diseases.
  2. History of any malignancy within the previous 5 years prior to Screening
  3. History of lymphoproliferative disease including lymphoma.
  4. History of congestive heart failure
  5. Physical incapacitation (ACR functional Class IV or wheelchair-/bed-bound).
  6. History of demyelinating disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Vencovsky, M.D., Ph.D., Principal Investigator — Charles University, Czech Republic
Locations (2):
- Investigational Site, Kielce, Poland
- Investigational Site, Southampton, Hampshire, United Kingdom

REFERENCES:
- [Derived] Emery P, Suh CH, Weinblatt ME, Smolen JS, Keystone EC, Genovese M, Vencovsky J, Kay J, Hong E, Baek Y, Ghil J. Impact of immunogenicity on efficacy and tolerability of tumour necrosis factor inhibitors: pooled analysis of biosimilar studies in rheumatoid arthritis. Scand J Rheumatol. 2020 Sep;49(5):361-370. doi: 10.1080/03009742.2020.1732458. Epub 2020 May 29. PMID 32468892
- [Derived] Smolen JS, Choe JY, Weinblatt ME, Emery P, Keystone E, Genovese MC, Myung G, Hong E, Baek I, Ghil J. Pooled analysis of TNF inhibitor biosimilar studies comparing radiographic progression by disease activity states in rheumatoid arthritis. RMD Open. 2020 Jan;6(1):e001096. doi: 10.1136/rmdopen-2019-001096. PMID 31958281
- [Derived] Emery P, Vencovsky J, Sylwestrzak A, Leszczynski P, Porawska W, Baranauskaite A, Tseluyko V, Zhdan VM, Stasiuk B, Milasiene R, Barrera Rodriguez AA, Cheong SY, Ghil J. 52-week results of the phase 3 randomized study comparing SB4 with reference etanercept in patients with active rheumatoid arthritis. Rheumatology (Oxford). 2017 Dec 1;56(12):2093-2101. doi: 10.1093/rheumatology/kex269. PMID 28968793
- [Derived] Emery P, Vencovsky J, Sylwestrzak A, Leszczynski P, Porawska W, Stasiuk B, Hilt J, Mosterova Z, Cheong SY, Ghil J. Long-term efficacy and safety in patients with rheumatoid arthritis continuing on SB4 or switching from reference etanercept to SB4. Ann Rheum Dis. 2017 Nov 13;76(12):1986-1991. doi: 10.1136/annrheumdis-2017-211591. PMID 28794078
- [Derived] Emery P, Vencovsky J, Sylwestrzak A, Leszczynski P, Porawska W, Baranauskaite A, Tseluyko V, Zhdan VM, Stasiuk B, Milasiene R, Barrera Rodriguez AA, Cheong SY, Ghil J. A phase III randomised, double-blind, parallel-group study comparing SB4 with etanercept reference product in patients with active rheumatoid arthritis despite methotrexate therapy. Ann Rheum Dis. 2017 Jan;76(1):51-57. doi: 10.1136/annrheumdis-2015-207588. Epub 2015 Jul 6. PMID 26150601

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SB4 (Proposed Biosimilar to Etanercept) | Enbrel (Etanercept)
Started | 299 | 297
Completed | 259 | 246
Not Completed | 40 | 51
Not completed — Adverse Event | 13 | 17
Not completed — Protocol Violation | 1 | 0
Not completed — Lack of Efficacy | 1 | 3
Not completed — Lost to Follow-up | 1 | 3
Not completed — Physician Decision | 15 | 10
Not completed — Withdrawal by Subject | 9 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SB4 (Proposed Biosimilar to Etanercept) | Enbrel (Etanercept) | Total
Number analyzed (Participants) | 299 | 297 | 596
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (11.72) | 51.6 (11.63) | 51.8 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 249 | 253 | 502
  Male | 50 | 44 | 94

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology 20% Response Criteria (ACR20)
Time Frame: Week 24
Measure: Number; unit: percentage of participants
Arm/Group | SB4 (Proposed Biosimilar to Etanercept) | Enbrel (Etanercept)
Number analyzed (Participants) | 247 | 236
percentage of participants | 78.1 | 80.5

2. Secondary Outcome: ACR20
Time Frame: Week 52
Measure: Number; unit: percentage of participants
Arm/Group | SB4 (Proposed Biosimilar to Etanercept) | Enbrel (Etanercept)
Number analyzed (Participants) | 224 | 216
percentage of participants | 80.8 | 81.5

3. Secondary Outcome: American College of Rheumatology 50% Response Criteria (ACR50)
Time Frame: Week 24, Week 52
Measure: Number; unit: percentage of participants
Groups:
- SB4 (Proposed Biosimilar to Etanercept) at Week 24; SB4 (Proposed Biosimilar to Etanercept) at Week 52: SB4 50 mg/week via subcutaneous injection
  SB4 (proposed biosimilar to etanercept)
- Enbrel (Etanercept) at Week 24; Enbrel (Etanercept) at Week 52: Enbrel 50 mg/week via subcutaneous injection
  Enbrel (etanercept)
Arm/Group | SB4 (Proposed Biosimilar to Etanercept) at Week 24 | Enbrel (Etanercept) at Week 24 | SB4 (Proposed Biosimilar to Etanercept) at Week 52 | Enbrel (Etanercept) at Week 52
Number analyzed (Participants) | 247 | 236 | 224 | 216
percentage of participants | 46.2 | 42.4 | 58.5 | 53.2

ADVERSE EVENTS:
Groups:
- SB4 (Proposed Biosimilar to Etanercept): SB4 50 mg/week via subcutaneous injection
  SB4 (proposed biosimilar to etanercept)
- Enbrel (Etanercept): Enbrel 50 mg/week via subcutaneous injection
  Enbrel (etanercept)
Arm/Group | SB4 (Proposed Biosimilar to Etanercept) | Enbrel (Etanercept)
Serious Adverse Events (participants affected / at risk) | 18/299 | 15/297
Other Adverse Events (participants affected / at risk) | 175/299 | 179/297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB4 (Proposed Biosimilar to Etanercept) (N=299) | Enbrel (Etanercept) (N=297)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary Failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1)
Chorioretinopathy (Eye disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Device Failure (General disorders) | 1 (1) | 0 (0)
Bile Duct Stone (Hepatobiliary disorders) | 1 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder Perforation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver Abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Still'S Disease Adult Onset (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine Polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal Prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB4 (Proposed Biosimilar to Etanercept) (N=299) | Enbrel (Etanercept) (N=297)
Leukopenia (Blood and lymphatic system disorders) | 6 (7) | 3 (4)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 5 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Anaemia Of Chronic Disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary Failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular Insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1)
Mitral Valve Prolapse (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
External Ear Inflammation (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 1 (1)
Thyroid Cyst (Endocrine disorders) | 0 (0) | 1 (1)
Eyelid Oedema (Eye disorders) | 2 (3) | 0 (0)
Conjunctival Haemorrhage (Eye disorders) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 1 (1) | 1 (1)
Eye Irritation (Eye disorders) | 1 (1) | 0 (0)
Eyelid Ptosis (Eye disorders) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Chorioretinopathy (Eye disorders) | 0 (0) | 1 (1)
Presbyopia (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 7 (8)
Abdominal Pain Upper (Gastrointestinal disorders) | 4 (5) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (8) | 1 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 4 (4)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum Intestinal (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocele (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Parotid Gland Inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 4 (5)
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2)
Portal Hypertensive Gastropathy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reflux Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Injection Site Erythema (General disorders) | 6 (16) | 33 (85)
Influenza Like Illness (General disorders) | 3 (5) | 1 (1)
Oedema Peripheral (General disorders) | 3 (3) | 3 (4)
Asthenia (General disorders) | 2 (2) | 5 (5)
Chest Pain (General disorders) | 2 (3) | 2 (3)
Chills (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 4 (4)
Injection Site Rash (General disorders) | 2 (2) | 6 (11)
Pain (General disorders) | 2 (2) | 1 (1)
Spinal Pain (General disorders) | 2 (3) | 1 (1)
Device Failure (General disorders) | 1 (1) | 0 (0)
Injection Site Haematoma (General disorders) | 1 (1) | 0 (0)
Injection Site Hypersensitivity (General disorders) | 1 (1) | 2 (10)
Injection Site Pruritus (General disorders) | 1 (1) | 4 (6)
Injection Site Reaction (General disorders) | 1 (1) | 8 (13)
Pyrexia (General disorders) | 1 (1) | 2 (3)
Application Site Erythema (General disorders) | 0 (0) | 3 (18)
Application Site Reaction (General disorders) | 0 (0) | 1 (1)
Face Oedema (General disorders) | 0 (0) | 1 (1)
Feeling Hot (General disorders) | 0 (0) | 1 (1)
Injection Site Bruising (General disorders) | 0 (0) | 1 (1)
Injection Site Dermatitis (General disorders) | 0 (0) | 1 (2)
Injection Site Inflammation (General disorders) | 0 (0) | 2 (2)
Injection Site Oedema (General disorders) | 0 (0) | 3 (6)
Injection Site Pain (General disorders) | 0 (0) | 1 (1)
Injection Site Swelling (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 2 (3)
Soft Tissue Inflammation (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 4 (4) | 0 (0)
Liver Disorder (Hepatobiliary disorders) | 3 (3) | 0 (0)
Cholecystitis Chronic (Hepatobiliary disorders) | 2 (3) | 0 (0)
Bile Duct Stone (Hepatobiliary disorders) | 1 (2) | 0 (0)
Biliary Colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder Perforation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergy To Arthropod Bite (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 24 (28) | 16 (18)
Nasopharyngitis (Infections and infestations) | 15 (17) | 16 (17)
Viral Infection (Infections and infestations) | 7 (7) | 5 (5)
Bronchitis (Infections and infestations) | 6 (6) | 6 (6)
Rhinitis (Infections and infestations) | 6 (6) | 4 (5)
Pharyngitis (Infections and infestations) | 5 (5) | 8 (9)
Urinary Tract Infection (Infections and infestations) | 5 (5) | 7 (9)
Oral Herpes (Infections and infestations) | 4 (7) | 5 (6)
Herpes Zoster (Infections and infestations) | 3 (5) | 1 (1)
Asymptomatic Bacteriuria (Infections and infestations) | 2 (3) | 0 (0)
Ear Infection (Infections and infestations) | 2 (2) | 0 (0)
Otitis Externa (Infections and infestations) | 2 (2) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 3 (3)
Acute Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Chronic Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 1 (1)
Fungal Infection (Infections and infestations) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Herpes Simplex (Infections and infestations) | 1 (1) | 2 (2)
Liver Abscess (Infections and infestations) | 1 (1) | 0 (0)
Localised Infection (Infections and infestations) | 1 (1) | 0 (0)
Lyme Disease (Infections and infestations) | 1 (1) | 0 (0)
Otitis Media (Infections and infestations) | 1 (1) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Rash Pustular (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Tinea Pedis (Infections and infestations) | 1 (1) | 1 (1)
Tinea Versicolour (Infections and infestations) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 2 (2)
Tooth Infection (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Acute Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Eczema Infected (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (2)
Herpes Virus Infection (Infections and infestations) | 0 (0) | 1 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Lobar Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Nail Candida (Infections and infestations) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pulpitis Dental (Infections and infestations) | 0 (0) | 1 (1)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Viral Rhinitis (Infections and infestations) | 0 (0) | 1 (2)
Vulvovaginal Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibula Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injection Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 18 (25) | 17 (26)
Aspartate Aminotransferase Increased (Investigations) | 8 (13) | 9 (10)
Gamma-Glutamyltransferase Increased (Investigations) | 5 (11) | 5 (6)
Lymphocyte Count Decreased (Investigations) | 4 (4) | 6 (8)
Transaminases Increased (Investigations) | 4 (5) | 4 (4)
Blood Pressure Increased (Investigations) | 3 (4) | 3 (3)
Liver Function Test Abnormal (Investigations) | 3 (4) | 2 (2)
Blood Alkaline Phosphatase Increased (Investigations) | 2 (4) | 0 (0)
Blood Glucose Increased (Investigations) | 2 (2) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 2 (4) | 0 (0)
Neutrophil Count Decreased (Investigations) | 2 (2) | 1 (1)
White Blood Cell Count Decreased (Investigations) | 2 (2) | 1 (1)
Blood Urine Present (Investigations) | 1 (1) | 0 (0)
Haemoglobin Decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil Count Increased (Investigations) | 1 (1) | 0 (0)
Nitrite Urine Present (Investigations) | 1 (1) | 0 (0)
Urine Analysis Abnormal (Investigations) | 1 (1) | 0 (0)
Weight Increased (Investigations) | 1 (1) | 0 (0)
Blood Calcium Decreased (Investigations) | 0 (0) | 1 (2)
Blood Phosphorus Decreased (Investigations) | 0 (0) | 2 (3)
Lymphocyte Count Abnormal (Investigations) | 0 (0) | 1 (1)
Lymphocyte Count Increased (Investigations) | 0 (0) | 1 (1)
Platelet Count Decreased (Investigations) | 0 (0) | 1 (3)
Platelet Count Increased (Investigations) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic Syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 9 (10) | 10 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (10)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fracture Delayed Union (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Sjogren'S Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Still'S Disease Adult Onset (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nuchal Rigidity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Periostitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal Deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma Of Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pyogenic Granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 13 (15) | 8 (16)
Dizziness (Nervous system disorders) | 2 (3) | 7 (7)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Anosmia (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance In Attention (Nervous system disorders) | 1 (1) | 0 (0)
Dystonia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 2 (3)
Stupor (Nervous system disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Balance Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Hypertensive Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Loss Of Consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Sleep Disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Initial Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Tachyphrenia (Psychiatric disorders) | 1 (1) | 0 (0)
Neurosis (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (3) | 2 (3)
Calculus Bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Tract Inflammation (Renal and urinary disorders) | 1 (1) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast Mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast Swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical Polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine Polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal Prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast Induration (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menopausal Symptoms (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 10 (11)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis Atrophic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (4)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Rash Papular (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4)
Erythema (Skin and subcutaneous tissue disorders) | 2 (4) | 10 (10)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema Annulare (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin Mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Umbilical Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Menopause (Social circumstances) | 0 (0) | 1 (1)
Tooth Extraction (Surgical and medical procedures) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 11 (16) | 11 (12)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least sixty (60) days prior to submitting or presenting a manuscript or other materials relating to the Study to a publisher, reviewer, or other outside persons, the Site shall provide to Sponsor a copy of all such manuscripts and materials, and allow Sponsor sixty (60) days to review and comment on them. If the Sponsor requests, the Site shall remove any Confidential Information (other than Study results) prior to submitting or presenting the materials.